CLINICAL TRIAL: NCT05252260
Title: Comparison Of Diode Laser-Assisted Vestibuloplasty And Conventional Vestibuloplasty In Terms Of Wound Healing And Vestibular Depth Gain
Brief Title: Comparison of Diode Laser-Assisted Vestibuloplasty And Conventional Vestibuloplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sadiye Gunpinar, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/120
Record Dates: First submitted 2022-02-02; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Wound Heal; Vestibular Abnormality; Low-level Light Therapy; Surgical Wound
MeSH Terms: conditions — Surgical Wound | interventions — Lasers, Semiconductor; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diode Laser (Experimental): Vestibuloplasty operation was performed via diode laser
  Interventions: Procedure: Diode Laser
- Diode laser + Low-level laser therapy (Other): Vestibuloplasty operation was performed via diode laser and following low-level laser therapy was applied
  Interventions: Procedure: Diode Laser; Other: Low level laser therapy (LLLT)
- Conventional surgery (Active Comparator): Vestibuloplasty operation was performed via scalpel
  Interventions: Procedure: Conventional Surgery
- Conventional surgery + Low-level laser therapy (Other): Vestibuloplasty operation was performed via scalpel and following low-level laser therapy was applied
  Interventions: Procedure: Conventional Surgery; Other: Low level laser therapy (LLLT)

INTERVENTIONS:
Procedure: Diode Laser — Vestibuloplasty surgery was performed via diode laser. Laser irradiation was performed in continuous wave mode, using a 980 nm diode laser with a power of 1.5W, 600 μm optical fiber.
  Arms: Diode Laser; Diode laser + Low-level laser therapy
Procedure: Conventional Surgery — A local anesthetic was administered bilaterally to the mental area and waited for 5 min for diffusion of the solution. Then, a horizontal incision was prepared at the mucogingival junction with a scalpel blade no. 15c. All the muscle fibers over the periosteum were resected carefully. Following, the mucosal flap was sutured to the depth of the vestibule sulcus with 4-0 polypropylene suture material, once every 4 mm, from a total of 5 regions.
  Arms: Conventional surgery; Conventional surgery + Low-level laser therapy
Other: Low level laser therapy (LLLT) — Vestibuloplasty surgery was performed via diode laser. Following, LLLT was applied in continuous wave mode for 1 minute without contacting the tissue, using a phototherapy probe (power output, 0.5W; total energy of 6 J / cm²) at a distance of 1-2 mm from the tissue. LLLT was repeated immediately after the surgery, on the 1st, 3rd and 7th days
  Arms: Conventional surgery + Low-level laser therapy; Diode laser + Low-level laser therapy

SUMMARY:
Randomized controlled parallel designed clinical study aimed to compare vestibule depth gain and dimensional changes of wound area in individuals who underwent vestibule deepening surgery using diode laser and conventional technique

DETAILED DESCRIPTION:
52 systemically healthy patients aged between 18 and 53 years (10 males and 42 females) with inadequate vestibular depth and insufficient attached gingiva in the anterior mandible were included in this randomized examiner- and patient-blinded, parallel design study. Following nonsurgical periodontal treatment, patients were divided into 4 groups as follows: a) diode laser (L); b) diode laser+Low level laser therapy (LLLT); c) conventional surgery and conventional surgery+LLLT, and vestibule deepening was applied to all subjects either with scalpel or laser assisted.

Scalpel surgery was performed as Clark's vestibuloplasty. A local anesthetic was administered bilaterally to the mental area. Then, a horizontal incision was prepared at the mucogingival junction with a scalpel blade 15c. All the muscle fibers over the periosteum were resected carefully. Following, the mucosal flap was sutured to the depth of the vestibule sulcus with 4-0 polypropylene suture material, once every 4 mm, from a total of 5 regions.

Laser assisted vestibuloplasty was performed using diode laser. Local anesthesia was achieved in the same manner as the control group (scalpel surgery). Laser irradiation was performed in continuous wave mode, using a 980 nm diode laser with a power of 1.5W, 600 μm optical fiber. After adequate local anesthesia, ablation was started from the mucogingival junction and performed with horizontal movements parallel to the bone. The muscle attachments were slowly released until the deepest point of the wound site was 5 mm. The mucosal flap was not stabilized with sutures and periodontal dressing was not used to cover the wound area.

ELIGIBILITY:
Inclusion Criteria:

* Patients were> 18 years old and of both genders,
* Patients presenting inadequate vestibular depth and insufficient attached gingiva on incisors in the mandibular anterior region
* Full mouth plaque index (PI) and gingival index (GI) scores < 1
* The patients had to be systemically healthy and nonsmokers

Exclusion Criteria:

* Patients who had Miller class II and more advanced gingival recession in the region of the lower anterior incisors and interproximal attachment loss
* Patients who were taking medications that would interfere with the wound-healing process, pregnant or lactating women,
* Patients who had previously undergone periodontal surgery in the study area, who had orthodontic therapy and using fixed/removable dentures involving lower anterior teeth were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Vestibule Depth Measurement Change (millimeter) | Change from Baseline vestibule depth measurement at 1 week; Change from Baseline vestibule depth measurement at 2 week; Change from Baseline vestibule depth measurement at 1 month
  Measurements were performed with the help of a plastic stopper placed on the endodontic canal instrument, with reference to the guides created on the acrylic stent which was prepared before the surgery

SECONDARY OUTCOMES:
Re-epithelization Area of the operation region | Change from baseline re-epithelization Area at 3 day; Change from baseline re-epithelization Area at 7 day; Change from baseline re-epithelization Area at 14 day
  Areas where there is little or no gingival epithelium were evaluated by applying a plaque staining agent to the surgical area. Clinical photographs of the stained gingiva were taken immediately after the operation and on the 3rd, 7th, and 14th days after the operation, using pre-prepared acrylic stents. Images were taken at standard magnification and distance on a digital camera (four optical zooms, 20cm) and the head of each patient was positioned to standardize the images. Incomplete epithelialized areas were measured using an image analysis software by the investigator blinded to the groups

OTHER OUTCOMES:
Wound Healing Scores of the surgical area | Wound healing scores on 3rd day, Wound healing scores on 7th day; Wound healing scores on 14th day; Wound healing scores on 28th day
  The healing of the surgical area was scored by using an index determined by Landry et al and compared between the groups in the evaluated time periods (1:worst and 5:excellent)
Pain and Loss of Function Scores of the study participants | Pain and Loss of Function on 1st day; Pain and Loss of Function on 7th day after the operation
  Patients were asked to rate their postoperative pain and functional changes (discomfort during eating and speaking) on visual analog scales (VAS) and compared between the groups in the evaluated time periods (1: minimum and 10: maximum). Minimum scores mean better results.
Change in horizontal wound dimension in the surgical area | Change from Baseline horizontal dimension at 1 week; Change from Baseline horizontal dimension at 2 week; Change from Baseline horizontal dimension at 4 week
  The linear dimensions of the wound in the horizontal direction were measured with a digital caliper over the projection on the endodontic file and recorded on the patient form.
Scar Tissue Formation Scores in the surgical area | Scar Tissue Formation at 1st month
  The scar tissue in the operation area was evaluated clinically and compared between the study groups (0: minimum scar formation; 8 maximum scar formation) minimum scar formation is better

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Gunpinar, Assoc. Prof, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Faculty of Dentistry, Department of Periodontology, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No